CLINICAL TRIAL: NCT02703558
Title: Evaluation of Fluorescein Use During Cystoscopy, a Randomized Control Trial
Brief Title: Evaluation of Fluorescein Use During Cystoscopy
Acronym: EFLUC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited interest from colleagues/time constraints
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00085778
Record Dates: First submitted 2016-02-26; First posted 2016-03-09 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Intraoperative Cystoscopy
MeSH Terms: interventions — Phenazopyridine; Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No dye (No Intervention): Participants will not receive a preoperative or intraoperative dye prior to their intraoperative concomitant cystoscopy.
- Phenazopyridine (Active Comparator): Participants will receive a single 200mg oral dose of phenazopyridine with a sip of water 30 minutes prior to their surgery which involves an intraoperative concomitant cystoscopy.
  Interventions: Drug: Phenazopyridine
- Fluorescein (Active Comparator): Participants will receive 0.25cc of 10% intravenous sodium fluorescein administered by anesthesia during their surgery, immediately prior to their intraoperative concomitant cystoscopy.
  Interventions: Drug: Fluorescein

INTERVENTIONS:
Drug: Phenazopyridine
  Other Names: Pyridium
  Arms: Phenazopyridine
Drug: Fluorescein
  Arms: Fluorescein

SUMMARY:
This study is a prospective randomized controlled study. Female patients over 18 years of age, who present for treatment of pelvic organ prolapse and/or stress urinary incontinence at the Pelvic Floor Center at the Johns Hopkins Bayview Medical Center, and who consent to undergo a urogynecologic surgical procedure, will be considered for inclusion in the study. Their histories will be reviewed by their attending surgeon and if they meet inclusion and exclusion criteria, they will be recruited for participation. The primary investigator and co-investigators (attending physician, fellows) will determine patient eligibility. Regarding privacy issues, the patients will be consented for both the procedure and for the study with careful attention made to emphasize patient confidentiality. When the patient presents for surgery, they will be randomized to receive either preoperative pyridium or intraoperative fluorescein or no dye. Given the color differences between the dyes, blinding will not occur. The process for recruitment will be consistent and any deviations from the protocol will be reported to the Johns Hopkins Internal Review Board.

ELIGIBILITY:
Inclusion Criteria:

• English speaking, female patients, ages 18 and older, undergoing urogynecologic surgery for pelvic organ prolapse or urinary incontinence with a planned concomitant cystoscopy at Johns Hopkins Bayview

Exclusion Criteria:

* Non-English speaking,
* Known allergic reactions or sensitivities to sodium fluorescein or phenazopyridine
* Known glucose-6-phosphate dehydrogenase or nicotinamide adenine dinucleotide- methemoglobin reductase deficiency
* Pregnant or breastfeeding
* Known renal disease or renal failure
* Undergoing concomitant non-urogynecologic procedures
* Dementia or cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Time required to complete cystoscopy | 30 min
  The attending surgeon of each case will document the time required to complete the cystoscopic assessment.
Time required to visualize ureteral jets | 30 min
  The attending surgeon of each case will document the time required to visualize the right and left ureters.

IPD SHARING:
Plan to Share IPD: No